CLINICAL TRIAL: NCT02694939
Title: Effectiveness of MI Enhanced Behavior Therapy for Adolescents With ADHD
Brief Title: STAND Community Trial
Acronym: STAND
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Florida International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: R01MH106587 (NIH)
Record Dates: First submitted 2015-07-24; First posted 2016-03-01 (Estimated); Last update posted 2021-02-03 (Actual); Status verified 2021-02

CONDITIONS: Attention Deficit Hyperactivity Disorder
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Behavior Therapy; Motivational Interviewing

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- STAND (Experimental): Receives STAND intervention delivered in community mental health setting.
  Interventions: Behavioral: STAND (Behavior Therapy + Motivational Interviewing)
- Usual Care (Active Comparator): Receives usual care from community therapists.
  Interventions: Behavioral: Usual Care

INTERVENTIONS:
Behavioral: STAND (Behavior Therapy + Motivational Interviewing) — Parent-teen collaborative skills based behavior therapy targeting Executive functioning and Delay Aversion in Teens
  Arms: STAND
Behavioral: Usual Care — Community Therapists free to deliver any therapy they feel is indicated.
  Arms: Usual Care

SUMMARY:
The proposed study evaluates the effectiveness of a family-based psychosocial treatment program for teens with ADHD (Supporting Teens' Academic Needs Daily; STAND) developed to be delivered in community settings. STAND is BT enhanced by Motivational Interviewing (MI) that was developed (R34 MH092466) for teens with ADHD through a stakeholder informed process. STAND consists of ten 50-minute sessions delivered by therapists with community-typical levels of training and supervision. Across randomized controlled pilot (N=28; N=36) and efficacy trials (N=128), STAND demonstrates medium to large effects on ADHD and ODD symptoms and indices of academic and family impairment. In the proposed study, 300 adolescents with ADHD who present for treatment at one of four community mental health agencies in Miami-Dade County, FL will be randomly assigned to STAND or agency usual care (UC). Participating agency therapists also will be randomly assigned to deliver STAND or UC. STAND therapists will receive a comprehensive treatment manual, three-day training, and weekly supervision from a project psychologist. Participants will be screened by research staff in the community setting and enrolled on a rolling basis over 30 months. Participants will be assessed at baseline, post-treatment, and three-month follow-up. In line with RDoC, multi-method measures will be obtained for treatment outcome (family and academic impairment), treatment mediators (executive functioning, parent academic involvement, parent-teen communication, parent/adolescent motivation, ADHD symptoms), and moderators of effectiveness (patient, practitioner, service delivery, and organization characteristics). Additional consumer perspective (satisfaction, therapeutic alliance) and agency fit (therapist competence, treatment fidelity, need for additional treatment, attendance, therapist attitude toward treatment, cost effectiveness) measures will also be obtained to evaluate effectiveness. We will recruit an ethnically diverse sample (65% Hispanic, 19% African-American, 16% Non-Hispanic White) that is historically underrepresented in research, but ideal for evaluating therapy effectiveness.

ELIGIBILITY:
Inclusion Criteria:

* ADHD diagnosis
* IQ of at least 70
* Enrollment in sixth through twelfth grade

Exclusion Criteria:

* history of autism spectrum disorder
* not attending a Miami-Dade County Public School
* a primary presenting problem other than ADHD, requiring immediate treatment of a different domain

Ages: 11 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 278 (Actual)
Dates: Start 2015-05 (Actual); Primary Completion 2018-12 (Actual); Study Completion 2020-10-31 (Actual)

PRIMARY OUTCOMES:
School Grades | 7 months
  GPA
ADHD Symptoms | 7 months
  Conners, ADHD Checklist
Behavior Problems in School | 7 months
  Official Disciplinary Records from School District
Academic Problems | 7 months
  Adolescent Academic Problems Checklist
Parent Teen Conflict | 7 months
  Conflict Behavior Questionnaire, Video Interaction Tasks

SECONDARY OUTCOMES:
Satisfaction with Treatment | 7 months
  Rating Scale of Patient Satisfaction with all aspects of Treatment
Quality of Therapeutic Relationship between the therapist and the patient | 7 months
  Patient report on therapeutic alliance
Organization Skills | 7 months
  Direct observation of recording homework and book bag organization
Executive Functioning | 7 months
  BRIEF rating scale, DKEFS, AWMA
Motivation | 7 months
  Motivation (readiness) ruler, hungry donkey task, choice delay task,
Parent academic Involvement | 7 months
  Parent report of academic management, number of hours spent helping, video interaction task
parent-teen communication | 7 months
  video tasks
parent readiness to change | 7 months
  Motivation (readiness) ruler, parent change talk

CONTACTS AND LOCATIONS:
Locations (1):
- Florida International University, Miami, Florida, United States

REFERENCES:
- [Derived] Sibley MH, Graziano PA, Coxe S, Page TF, Martin P. Three-Year Effects of Motivational Interviewing-Enhanced Behavior Therapy for Adolescents With Attention-Deficit/Hyperactivity Disorder: A Randomized Community-Based Trial. J Am Acad Child Adolesc Psychiatry. 2025 Oct;64(10):1165-1178. doi: 10.1016/j.jaac.2024.10.009. Epub 2024 Oct 21. PMID 39442667
- [Derived] Sibley MH, Ortiz M, Rios-Davis A, Zulauf-McCurdy CA, Graziano PA, Bickman L. Stakeholder-Generated Implementation Strategies to Promote Evidence-Based ADHD Treatment in Community Mental Health. Adm Policy Ment Health. 2022 Jan;49(1):44-58. doi: 10.1007/s10488-021-01143-5. Epub 2021 May 14. PMID 33988847
- [Derived] Sibley MH, Graziano PA, Coxe S, Bickman L, Martin P. Effectiveness of Motivational Interviewing-Enhanced Behavior Therapy for Adolescents With Attention-Deficit/Hyperactivity Disorder: A Randomized Community-Based Trial. J Am Acad Child Adolesc Psychiatry. 2021 Jun;60(6):745-756. doi: 10.1016/j.jaac.2020.07.907. Epub 2020 Aug 28. PMID 32861773
- [Derived] Sibley MH, Graziano PA, Bickman L, Coxe SJ, Martin P, Rodriguez LM, Fallah N, Ortiz M. Implementing Parent-Teen Motivational Interviewing + Behavior Therapy for ADHD in Community Mental Health. Prev Sci. 2021 Aug;22(6):701-711. doi: 10.1007/s11121-020-01105-7. PMID 32103410